CLINICAL TRIAL: NCT00841841
Title: Dipyrone Versus Acetaminophen in the Control of Postoperative Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Center of Araraquara (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Thallita Pereira Queiroz, Thallita Pereira Queiroz, DDS, MSc, PhD, University Center of Araraquara
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: upeclin/FOA-Unesp-02
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Pain, Postoperative
Keywords: Analgesia; molar third; acetaminophen; dipyrone
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Dipyrone; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dipyrone (Experimental): Analgesic affectiveness using Dipyrone (500mg) as a postoperative drug for pain relief.
  Intervention: "Drug: dipyrone and acetaminophen"
  Interventions: Drug: dipyrone and acetaminophen
- Acetaminophen (Experimental): Analgesic affectiveness using Acetaminophen (750mg) as a postoperative drug for pain relief.
  Intervention: "Drug: dipyrone and acetaminophen"
  Interventions: Drug: dipyrone and acetaminophen

INTERVENTIONS:
Drug: dipyrone and acetaminophen — The patients were randomly assigned to 2 groups of 15 patients, according to the drug prescribed as postoperative medication: Group I: dipyrone 500 mg every 6 hours (4 males, 11 females, mean age = 25.2 years) and Group II: paracetamol 750 mg every 6 hours (3 males, 12 females, mean age = 26.8 years)
  Other Names: Dipyrone: Novalgina; Acetaminophen: Tylenol

SUMMARY:
Adequate postoperative pain management is challenging for practitioners despite recent advances in pain control techniques and analgesic agents. The purpose of this study is to compare the efficacy of Dipyrone and acetaminophen in postoperative pain after third molar surgery.

DETAILED DESCRIPTION:
Thirty patients scheduled for surgical removal of impacted third molars at the Discipline of Oral and Maxillofacial Surgery and Traumatology of the Dental School of Araçatuba, São Paulo State University, Brazil, were selected for the study after review and approval of the research protocol by the institutional Research Ethics Committee (Protocol #2006-01083). All patients received verbal and written explanations about the study purposes and procedures, and all of them signed an informed consent form prior to enrollment.

Patients should be in good general health and those who fulfilled any of the following criteria were excluded: systemic disorders; known hypersensitivity to any of the study medications; pregnancy or nursing; local contraindication to surgery as judged by the oral surgeon; and use of any analgesic agent 24 hours before surgery.

All patients were premedicated with oral dexamethasone 4 mg one hour before surgery for modulation of the postoperative edema. The surgical procedures were performed by a single operator according to a standardized surgical protocol and in compliance with all principles of the surgical technique. All patients received standard verbal and written postoperative instructions regarding diet, oral hygiene and general care.

The patients were randomly assigned to 2 groups of 15 patients, according to the drug prescribed as postoperative medication: Group I: dipyrone 500 mg every 6 hours (4 males, 11 females, mean age = 25.2 years) and Group II: paracetamol 750 mg every 6 hours (3 males, 12 females, mean age = 26.8 years). Amoxicillin 500 mg was prescribed for all patients. All surgeries were completed within 1 hour and were performed under local anesthesia with injection of an average volume of 3.6 mL of 2% mepivacaine with 1:100,000 adrenaline per surgical site. No relevant perioperative complications were observed.

In Group I, 3 maxillary right third molars, 9 maxillary left third molars, 10 mandibular left third molars and 9 mandibular right third molars were extracted. The following impaction positions were observed: vertical (n=22), horizontal (n=4) and medio-angulated (n=4). During surgery, osteotomy was necessary in 2 surgical sites and osteotomy associated with tooth sectioning was required in 8 cases. In Group II, 1 maxillary right third molar, 9 maxillary left third molars, 12 mandibular left third molar and 3 mandibular right third molars were extracted. The following impaction positions were observed: vertical (n=18), horizontal (n=2) and medio-angulated (n=3). During surgery, osteotomy, tooth sectioning and osteotomy associated with tooth sectioning were performed in 6, 3 and 6 cases, respectively.

Pain intensity was rated by the patients using a 4-point visual analog scale (VAS): 0 (no pain), 1 (mild pain), 2 (moderate pain), 3 (severe pain), 4 (unendurable pain). Measurements of pain intensity were performed in the immediate postoperative period and every 6 hours after surgery until completing 48 hours. Reports on the relief of the different pain intensities were obtained from the patients at the pre-established intervals (6 hours) using an ordinal scale in order to obtain the mean pain intensity scores for each patient and for each group. The use of a nonparametric statistical test was thus required for data comparison. Mann-Whitney test was used to compare the study groups by analyzing the mean pain intensity scores obtained every 6 hours, in the first 24 hours, in the final 24 hours and in the total 48-hour period. Significance level was set at 5%

ELIGIBILITY:
Inclusion Criteria:

* good general health

Exclusion Criteria:

* systemic disorders; known hypersensitivity to any of the study medications; pregnancy or nursing; local contraindication to surgery as judged by the oral surgeon; and use of any analgesic agent 24 hours before surgery.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2006-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Pain control with analgesics drugs | forty-eight hours

SECONDARY OUTCOMES:
visual analog scale | forty-eight hours

CONTACTS AND LOCATIONS:
Overall Officials: Thallita P Queiroz, MSc, Principal Investigator — São Paulo State University - UNESP